CLINICAL TRIAL: NCT00569179
Title: A PHASE I TRIAL OF ALLOREACTIVE NK CELLS INFUSION FOLLOWING TRANSPLANTATION OF HAPLOTYPE MISMATCHED, KIR MISMATCHED HIGHLY PURIFIED CD34 CELLS IN PATIENTS WITH ADVANCED OR REFRACTORY MYELOID MALIGNANCIES
Brief Title: A Phase I Trial of Alloreactive Cell Infusion Following Transplantation of Haplotype Cells in Patients With Myeloid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0612-26/ IUCRO-0179
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Lymphoid; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic
Keywords: Myeloid Malignancies; Bone Marrow Transplant; AML; ALL; MDS; CML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Lymphoid; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alloreactive NK cell infusion (Experimental): Escalating doses of alloreactive NK cells.
  Interventions: Device: CliniMACS CD34 Reagent System

INTERVENTIONS:
Device: CliniMACS CD34 Reagent System — Alloreactive NK cells will be purified by a two-step immunomagnetic selection (CD3 depletion followed by CD56 selection) using the CliniMACS device.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of alloreactive NK cells that can be transfused following stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented AML, ALL, MDS, CML,
* Identification of haploidentical donor
* LVEF > 45% corrected
* DLCO > 50% predicted
* Serum Creatinine <= 2 mg/dL
* Bilirubin < 2 x ULN
* AST, ALT < 2 x ULN
* Age ≤ 65 years
* Performance Status 0-1

Exclusion Criteria:

* Patients relapsing <6 months after autologous SCT are not eligible.
* Patients with active infections requiring oral or intravenous antibiotics are not eligible for enrollment until resolution of infection
* No HIV disease
* Non-pregnant and non-nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-08; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Investigate the maximum-tolerated dose (MTD) of highly-purified alloreactive NK cells infused following haplotype-mismatched, KIR ligand-mismatched transplants in patients with refractory hematological malignancies. | through Day 128

SECONDARY OUTCOMES:
Assess toxicity associated with the infusion of alloreactive NK cells | through Day 128
Assess the risk of acute and chronic GvHD following infusion of alloreactive NK cells. | through Day 128
Assess the feasibility of multiple harvesting and purifying NK cells to the relatively high-doses. | through Day 128
Describe the frequency and type of infections occurring within the first year following transplantation. | through Day 128
Describe immune reconstitution following transplantation. | through Day 128

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Farag, MD, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States